CLINICAL TRIAL: NCT05971433
Title: Determining the Role of Sympathetic Activity in the Impact of Combat Injury on Sleep and Cardiovascular Outcomes (SPIRIT)
Brief Title: Sympathetic Activity in Post-injury Outcomes: Impact on Sleep and caRdiovascular Health InvesTigation
Acronym: SPIRIT
Status: Enrolling by invitation | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Naval Health Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ian Stewart, Professor of Medicine; Director, Division of Nephrology, Uniformed Services University of the Health Sciences
Other Study IDs: USUHS.2022-110
Record Dates: First submitted 2023-06-27; First posted 2023-08-02 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Cardiovascular Diseases; Sleep Disorder; Arrythmia; Sympathetic Nervous System; Injury Traumatic
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Sleep Wake Disorders; Arrhythmias, Cardiac; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Injury severity scored as "severe": This group will include participants whose injury was scored as "severe" based on the recorded Injury Severity Score (ISS). Both cohorts will complete the same course of testing in this study.
- Injury severity scored as "minimal": This group will include participants whose injury was scored as "minimal" based on the recorded Injury Severity Score (ISS). Both cohorts will complete the same course of testing in this study.

SUMMARY:
The goal of this observational study is to learn about the long-term health of United States military service members who were injured during combat. The main questions it aims to examine are:

* How does the severity of a combat injury impact 1) cardiovascular risk, 2) the sympathetic nervous system and arrhythmias, 3) blood pressure, and 4) sleep disorders?
* Are self-reported mental health symptoms related to sympathetic nervous system hyperactivity, sleep disorders, and cardiovascular risk in combat-injured service members?

This study will recruit from a sample of participants in another research study called the Wounded Warrior Recovery Project (WWRP) who 1) agreed to be contacted about future research studies and 2) have a record of a combat injury within the Injury Severity Score ranges required for this study.

Participants will:

* Provide demographic information and a medical history review
* Visit a local laboratory for biometrics measurements and to provide blood and urine samples
* Wear an ambulatory electrocardiogram monitor for 24 hours per day for seven consecutive days
* Wear a home sleep test monitoring device for one night
* Wear a blood pressure monitor for 24 consecutive hours on the day after the home sleep test

At the end of the study, participants will be asked to mail back the home sleep test and blood pressure monitors. Prepaid package materials will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Wounded Warrior Recovery Project (WWRP) and previously agreed to be contacted regarding future research
* Able to complete the informed consent process, be mailed study devices, and complete laboratory draws within the United States
* Age greater than or equal to 18 years

Exclusion Criteria:

* No Injury Severity Score or 3 < Injury Severity Score < 15
* Unable to complete the informed consent process, be mailed study devices, and complete laboratory draws within the United States
* Not enrolled in the WWRP or enrolled in the WWRP but did not agree to be contacted about future research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wounded Warrior Recovery Project participants who 1) agreed to be contacted about future research studies and 2) have a record of injury within the established Injury Severity Score cutoffs for this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of arrhythmias | 7 days of wear
  Readings from a 24-hour ambulatory electrocardiogram (ECG) monitor will be used to determine the frequency of arrhythmias.
Frequency of atrial fibrillation | 7 days of wear
  Readings from a 24-hour ambulatory electrocardiogram (ECG) monitor will be used to determine the frequency of atrial fibrillation.
Frequency of atrial flutter | 7 days of wear
  Readings from a 24-hour ambulatory electrocardiogram (ECG) monitor will be used to determine the frequency of atrial flutter.
Density of premature ventricular contractions (PVCs) | 7 days of wear
  Readings from a 24-hour ambulatory electrocardiogram (ECG) monitor will be used to determine the density of PVCs (percentage of total heartbeats that are PVCs).
Frequency of ventricular tachycardia | 7 days of wear
  Readings from a 24-hour ambulatory electrocardiogram (ECG) monitor will be used to determine the frequency of ventricular tachycardia.
Heart rate | 7 days of wear
  Readings from a 24-hour ambulatory electrocardiogram (ECG) monitor will be used to determine heart rate.
Standard deviation of beat-to-beat intervals (SDNN) | 7 days of wear
  Standard deviation of beat-to-beat intervals (SDNN) is a heart rate variability (HRV) time domain measure that will be automatically calculated for each 5-min epoch of the 24-hour ambulatory electrocardiogram (ECG) recording.
Root mean square of successive differences (RMSSD) | 7 days of wear
  Root mean square of successive differences (RMSSD) is a heart rate variability (HRV) time domain measure that will be automatically calculated for each 5-min epoch of the 24-hour ambulatory electrocardiogram (ECG) recording.
Low frequency power | 7 days of wear
  Low frequency power (LF, 0.04 - 0.15 Hz) is a heart rate variability (HRV) frequency domain measure that will be automatically calculated for each 5-min epoch of the 24-hour ambulatory electrocardiogram (ECG) recording.
High frequency power | 7 days of wear
  High frequency power (HF, 0.15 - 0.4 Hz) is a heart rate variability (HRV) frequency domain measure that will be automatically calculated for each 5-min epoch of the 24-hour ambulatory electrocardiogram (ECG) recording.
Log-transformed QT variance (logQTv) | 7 days of wear
  Log-transformed QT variance (logQTv) s a QT variability (QTV) measure that will be automatically calculated for each 5-min epoch of the 24-hour ambulatory electrocardiogram (ECG) recording.
Beat-to-beat QT variability index (QTVI) | 7 days of wear
  Beat-to-beat QT variability index (QTVI) is a QT variability (QTV) measure that will be automatically calculated for each 5-min epoch of the 24-hour ambulatory electrocardiogram (ECG) recording.
Presence of obstructive sleep apnea | One night
  The presence of comorbid obstructive sleep apnea and/or nocturnal hypoxemia, will be evaluated with a home sleep study test device (HST) worn during the second or third study day
Presence of nocturnal hypoxemia | One night
  The presence of comorbid obstructive sleep apnea and/or nocturnal hypoxemia, will be evaluated with a home sleep study test device (HST) worn during the second or third study day
24-hour ambulatory blood pressure monitor (ABPM) | 24 hours
  Blood pressure (diastolic and systolic) will be assessed using a 24-hour ABPM worn during the 24-hour period following the HST.
High sensitivity C-reactive protein (hs-CRP) | Baseline
  This inflammatory marker will be measured during laboratory testing.
Posttraumatic Stress Disorder Checklist for Diagnostic and Statistics Manual of Mental Disorder 5 (PCL-5) | Baseline
  The severity of Posttraumatic Stress Disorder (PTSD) symptoms will be assessed by the PCL-5 20-question survey. Total scores range from 0 - 80, with higher scores indicating greater PTSD symptom severity.
8-item Patient Health Questionnaire depression scale (PHQ-8) | Baseline
  The severity of depressive symptoms will be measured by the eight-question PHQ-8 survey. Total scores range from 0 - 24, with with higher scores indicating greater depressive symptom severity.
Brief Dissociative Experience Scale (DES-B) | Baseline
  Severity of dissociative experiences will be assessed using the 8-item DES-B survey. Total scores range from 0 - 32, with with higher scores indicating greater dissociative experience severity.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  Participant-reported sleep characteristics will be assessed using the 19-item Pittsburgh Sleep Quality Index (PSQI). Total scores range from 0 - 21, with higher scores indicating worse sleep quality.
Epworth Sleepiness Scale (ESS) | Baseline
  Participant-reported sleep characteristics will be assessed using the 8-item Epworth Sleepiness Scale (ESS). Total scores range from 0 - 24, with higher scores indicating increased daytime sleepiness.
Insomnia Severity Index (ISI) | Baseline
  Participant-reported sleep characteristics will be assessed using the 7-item Insomnia Severity Index (ISI). Total scores range from 0 - 28, with higher scores indicating increased insomnia symptoms.
Berlin Sleep Questionnaire | Baseline
  Participant-reported sleep characteristics will be assessed using the 11-item Berlin Sleep Questionnaire. Scores will be calculated to determine if participants are "High Risk" or "Low Risk" for sleep apnea.
Body Mass Index | Baseline
  Height and weight will be measured during laboratory visit and combined to report BMI in kg/m^2.
Blood Pressure | Baseline
  Blood pressure (diastolic and systolic) will be recorded at the time of laboratory visit
Hemoglobin A1C (HBA1C) | Baseline
  This laboratory test will be used to assess overall health outcomes.
Alanine aminotransferase (ALT/SGPT) | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Albumin:globulin (A:G) ratio | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Albumin, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Alkaline phosphatase, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Aspartate aminotransferase (AST/SGOT) | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Bilirubin, total | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Blood urea nitrogen (BUN) | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Blood urea nitrogen (BUN):creatinine ratio | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Calcium, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Carbon dioxide, total | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Chloride, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Creatinine, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Estimated glomerular filtration rate (eGFR) calculation | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Globulin, total | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Glucose, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Potassium, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Protein, total, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Sodium, serum | Baseline
  This laboratory test will be measured as part of a comprehensive metabolic panel and will be used to assess overall health outcomes.
Cystatin C with estimated glomerular filtration rate (eGFR) | Baseline
  This laboratory test will be used to assess overall health outcomes.
Cholesterol, total | Baseline
  This laboratory test will be measured as part of a lipid panel and will be used to assess overall health outcomes.
High-density lipoprotein (HDL) cholesterol | Baseline
  This laboratory test will be measured as part of a lipid panel and will be used to assess overall health outcomes.
Low-density lipoprotein (LDL) cholesterol (calculation) | Baseline
  This laboratory test will be measured as part of a lipid panel and will be used to assess overall health outcomes.
Triglycerides | Baseline
  This laboratory test will be measured as part of a lipid panel and will be used to assess overall health outcomes.
Very low-density lipoprotein (VLDL) cholesterol (calculation) | Baseline
  This laboratory test will be measured as part of a lipid panel and will be used to assess overall health outcomes.
Albumin/creatinine ratio, random urine | Baseline
  This laboratory test will be used to assess overall health outcomes.
N-terminal pro b-type natriuretic peptide (NT-proBNP) | Baseline
  This laboratory test will be used to assess overall health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stewart, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walker LE, Jurick SM, Thomas V, Arnold T, Elisman K, Kalra S, Mains A, Rioux S, Galarneau M, McCabe C, Lavender JM, Collen J, Haigney MC, Solhjoo S, Stewart IJ. A study protocol for determining the role of Sympathetic activity in Post-injury outcomes: Impact on sleep and caRdiovascular health InvesTigation (SPIRIT). PLoS One. 2025 Jul 17;20(7):e0321035. doi: 10.1371/journal.pone.0321035. eCollection 2025. PMID 40674309